CLINICAL TRIAL: NCT02893397
Title: Pre-Surgical Supervised Exercise for Bone Cancer Patients
Brief Title: Supervised Exercise in Improving Physical Fitness Before Surgery in Patients With Resectable Bone Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Purpose: Supportive Care
Other Study IDs: 2016-0411; NCI-2016-01969 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0411 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-08-31; First posted 2016-09-08 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Malignant Bone Neoplasm
MeSH Terms: conditions — Bone Neoplasms | interventions — Fitness Trackers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (supervised exercise) (Experimental): Patients wear a fitbit and undergo supervised physical therapy exercise sessions over 40 minutes 3-5 times a week for at least 4 weeks.
  Interventions: Behavioral: Exercise Intervention
- Group II (fitbit) (Experimental): Patients wear a fitbit.
  Interventions: Device: Activity Monitor

INTERVENTIONS:
Device: Activity Monitor — Wear a fitbit
  Other Names: Activity Tracker; Activity Tracker Device; Physical Activity Measuring Device
  Arms: Group II (fitbit)
Behavioral: Exercise Intervention — Undergo supervised exercise sessions
  Arms: Group I (supervised exercise)

SUMMARY:
This clinical trial studies how well supervised exercise works in improving physical fitness before surgery in patients with bone cancer that can be removed by surgery. Supervised exercise may provide better short-term physical fitness in patients with bone cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if regular exercise, which may improve delivery and efficacy of chemotherapy, is feasible in children and young adults with malignant bone tumors undergoing neoadjuvant chemotherapy.

SECONDARY OBJECTIVES:

I. To determine if exercise results in a change in tumor vascularity as evidenced by magnetic resonance imaging (MRI) in children and young adults with malignant bone tumors who participate in structured aerobic exercise as compared to children and young adults who do not.

II. To determine whether serum levels of thrombospondin-1, an endogenous anti-angiogenic protein, and sphingosine-1-phosphate, an angiogenic modulator, increase in children and young adults with malignant bone tumors who participate in supervised aerobic exercise over a 4 week period of time during neoadjuvant chemotherapy.

III. To determine if aerobic exercise decreases reactive oxygen species (ROS) in the peripheral blood of bone sarcoma patients.

IV. To determine if the numbers of circulating tumor cells decrease in patients who participate in supervised exercise over a 4 week period of time.

V. To determine whether a home-based exercise program or supervised exercise program is more feasible for this patient population.

OUTLINE: Patients are assigned to 1 of 2 groups.

GROUP I: Patients wear a fitbit and undergo supervised physical therapy exercise sessions over 40 minutes 3-5 times a week for at least 4 weeks.

GROUP II: Patients wear a fitbit.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a new diagnosis of primary bone tumor, and whose treatment plan includes surgery
* Patients who are expected to receive at least 4 weeks of neoadjuvant chemotherapy treatment between enrollment in the study and planned surgery
* Participants willing to wear a Fitbit

Exclusion Criteria:

* Patients who are not receiving their primary cancer care (surgery and chemotherapy) at MD Anderson Cancer Center (participants from the supervised exercise group only)
* Patients who have a cognitive disorder which impacts the ability to follow directions or adhere to safety rules; this will be determined by the physical therapist by assessing whether a neurological disorder or musculoskeletal disorder would prevent the patient from safely exercising
* Patients who have a neurological or structural disorder which would impact use of exercise equipment; this will be determined by the physical therapist by assessing whether a neurological disorder or musculoskeletal disorder would prevent the patient from safely exercising
* Any patient who, in the opinion of the investigators, will be unable to comply with a supervised exercise regimen
* Any concurrent co-morbid illness and/or infection which in the opinion of the investigators could make the patient unable to comply fully with the trial procedures

Ages: 5 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2016-08-30 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility defined as at least 10 of out 15 patients in the supervised exercise group complete more than or equal to 75% (9 of 12 sessions) supervised physical therapy exercise sessions | At least 4 weeks
  Completion of daily exercise is defined as at least 20 minutes of aerobic exercise achieved within heart rate and blood pressure that the licensed physical therapist has determined is safe for the patient on that given day.

SECONDARY OUTCOMES:
Change in tumor vascularity as measured by magnetic resonance imaging diffusion studies | Baseline up to 4 weeks
  Will use a two-sided t-test with a significance level of 5% to compare the tumor vascularity between groups.
Change in tumor vascularity as measured by blood serum analysis of serum thrombospondin-1 and sphingosine-1-phosphate | Baseline up to 4 weeks
  Will use a two-sided t-test with a significance level of 5% to compare the tumor vascularity between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Valerae O Lewis, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - M D Anderson Cancer Center, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org